CLINICAL TRIAL: NCT03629353
Title: The Efficacy of Transnasal Humidified Rapid-insufflation Ventilatory Exchange in Patients Undergoing Laryngeal Microsurgery: a Randomized Controlled Trial
Brief Title: The Efficacy of Transnasal Humidified Rapid-insufflation Ventilatory Exchange During Laryngeal Microsurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THRIVE during LMS
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2018-09

CONDITIONS: Apneic Oxygenation
Keywords: airway management; high flow nasal cannula; laryngeal microsurgery
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intubation group (Experimental): The enrolled patients will be oxygenated by endotracheal tube during operation.
  Interventions: Procedure: endotracheal intubation
- THRIVE group (Experimental): The enrolled patients will be oxygenated by intubationless high flow nasal cannula during operation.
  Interventions: Procedure: high flow nasal cannula

INTERVENTIONS:
Procedure: endotracheal intubation — After preoxygenation with FiO2 1.0 and flow rate of 8 L/min for 3 minutes, the enrolled patients will be intubated with endotracheal tube and maintained oxygenation during surgery.
  Arms: intubation group
Procedure: high flow nasal cannula — After preoxygenation with 100% oxygen through high flow nasal cannula for 3 minutes, the enrolled patients will be maintained intubationless oxygenation with flow rate of 70 L/min during surgery.
  Arms: THRIVE group

SUMMARY:
Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) was revealed to prolong apneic time with a slow increase in carbon dioxide; thus, has been used for preoxygenation in patients with difficult airways or requiring rapid sequence induction in general anesthesia.

However, in patients undergoing hypopharyngeal and laryngo-tracheal surgery, THRIVE during operation can be advantageous by allowing tubeless surgical field with sufficient oxygenation.

Therefore, the investigators conducted this study to evaluate the efficacy of THRIVE on prolonged apneic time with enhanced surgical conditions in patients with laryngeal microsurgery.

DETAILED DESCRIPTION:
Patients undergoing laryngeal microsurgery will be randomized into either intubation group or THRIVE group.

On arriving operating room, the patients will be preoxygenated by facemask or high flow nasal cannula with 100% oxygen for 3 minutes according to the allocated group. After inducing general anesthesia, patients in intubation group will be oxygenated by endotracheal tube, while patients in THRIVE group will be oxygenated by high flow nasal cannula with flow rate of 70L/min. During the surgery, the endotracheal tube can be removed and reintubated in intubation group patients to provide surgical field by a surgeon, respectively.

The monitored pulse oximetry, oxygen reserve index, and transcutaneous partial pressure of carbon dioxide will be recorded during surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laryngeal microsurgery
* ASA class I-III

Exclusion Criteria:

* patients scheduled for laryngeal microsurgery using CO2 laser
* patients with increased intracranial pressure
* patients with skull base defect
* patients with chronic obstructive pulmonary disease
* patients with pulmonary hypertension
* patients requiring rapid sequence induction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
lowest oxygen saturation | from the time of starting laryngeal microsurgery till the end of the surgery
  lowest oxygen saturation monitored by pulse oximetry during laryngeal microsurgery

SECONDARY OUTCOMES:
lowest oxygen reserve index | from the time of starting laryngeal microsurgery till the end of the surgery
  lowest oxygen reserve index monitored during laryngeal microsurgery
highest transcutaneous partial pressure of carbon dioxide | from the time of starting laryngeal microsurgery till the end of the surgery
  highest transcutaneous partial pressure of carbon dioxide monitored during laryngeal microsurgery

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Min SH, Yoon H, Huh G, Kwon SK, Seo JH, Cho YJ. Efficacy of high-flow nasal oxygenation compared with tracheal intubation for oxygenation during laryngeal microsurgery: a randomised non-inferiority study. Br J Anaesth. 2022 Jan;128(1):207-213. doi: 10.1016/j.bja.2021.09.016. Epub 2021 Oct 20. PMID 34688473